CLINICAL TRIAL: NCT01051999
Title: Glutamine Supplementation and Immunity in Adults With Cystic Fibrosis
Brief Title: Glutamine Supplementation in Cystic Fibrosis
Acronym: CFG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Emmaus Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Thomas R. Ziegler, MD, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00025564
Record Dates: First submitted 2010-01-15; First posted 2010-01-20 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Cystic Fibrosis; Immune Function
Keywords: Glutamine
MeSH Terms: conditions — Cystic Fibrosis | interventions — Glutamine; Alanine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glutamine (Experimental): Patients randomized to the glutamine arm will receive 0.7g/kg of oral glutamine powder per day
  Interventions: Dietary Supplement: Glutamine
- Placebo (Placebo Comparator): Patients randomized to the placebo arm will receive 0.7g/kg of oral isonitrogenous L-alanine powder per day
  Interventions: Dietary Supplement: L-alanine

INTERVENTIONS:
Dietary Supplement: Glutamine — Oral glutamine powder
  Arms: Glutamine
Dietary Supplement: L-alanine — L-alanine oral powder
  Arms: Placebo

SUMMARY:
Patients with cystic fibrosis develop frequent and potentially life-threatening lung infections. Recent studies suggest that the nutrient "glutamine" may help the body fight off infection. Glutamine is an amino acid; a type of nutrient the body requires to build muscle. It is one of the building blocks of protein. During an illness, blood levels of glutamine tend to be lower than normal. Also, many patients with cystic fibrosis have difficulty getting normal levels of nutrients from food. The aim of this study is to see if patients with cystic fibrosis have low levels of glutamine when they experience an infection, and whether a dietary glutamine supplement taken daily for three months can raise these levels. We also want to see if this supplement can improve other blood markers of immunity (the body's ability to defend itself from infection). We hope to enroll 40 people with cystic fibrosis who experience a lung infection, over a one year period, into this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years of age) with cystic fibrosis who give informed consent
* Patients must have a clinically diagnosed pulmonary exacerbation at time of enrollment, characterized by clinical requirement for oral or intravenous antibiotics associated with pulmonary symptoms such as increased cough or decreased forced expiratory volumes (FEV1)
* Participants must agree to provide phlebotomy samples and complete all study protocol at presentation and at return visits

Exclusion Criteria:

* Any patients taking specific glutamine supplements within 30 days of enrollment
* Pregnant or lactating women
* Patients involved in any other research protocol involving intake of a study drug, in the last 60 days.
* Patients who are chronically immunosuppressed due to drugs or immunosuppressive illness other than CF (e.g. HIV/AIDS, chronic autoimmune disease)
* Patients receiving hemodialysis or with creatinine >2.5mg/dL
* Patients with liver failure from any cause
* Patients with a history of cancer within the past 12 months or currently receiving anti-neoplastic therapy.
* Patients with a history of seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Percent increase in plasma glutamine and glutathione redox levels measured at weeks 0, 4, 8, and 12. | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Atlanta, Georgia, United States